CLINICAL TRIAL: NCT01890200
Title: A Phase III, Randomized, Double Blind, Placebo Controlled Study to Evaluate the Effects of Adding TCM-700C,Botanical Drug, on the Standard Treatment (Peginterferon and Ribavirin) for Subjects With Naive Genotype 1 Hepatitis C Infection
Brief Title: The Effects of Adding TCM-700C on the Standard Combination Treatment for HCV Genotype 1 Patients(Phase III)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: TCM Biotech International Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCM-700-02-01
Record Dates: First submitted 2013-06-26; First posted 2013-07-01 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2016-01

CONDITIONS: Chronic Hepatitis C
Keywords: add-on treatment; botanical drug; HCV genotype 1; TCM-700C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TCM-700C (low dose) (Experimental): an add-on drug (t.i.d) to conventional treatment(Peginterferon alfa-2a + ribavirin) of Hepatitis C
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin; Drug: TCM-700C
- TCM-700C (high dose) (Experimental): an add-on drug (t.i.d) to conventional treatment(Peginterferon alfa-2a + ribavirin) of Hepatitis C
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin; Drug: TCM-700C
- Placebo (Placebo Comparator): placebo add on(t.i.d) to conventional treatment(Peginterferon alfa-2a + ribavirin) of Hepatitis C
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin; Drug: Placebo

INTERVENTIONS:
Drug: Peginterferon alfa-2a — conventional treatment of Hepatitis C
  Other Names: Pegasys
Drug: Ribavirin — conventional treatment of Hepatitis C
  Other Names: Rebetol
Drug: TCM-700C — An add-on drug to conventional treatment of Hepatitis C
  Arms: TCM-700C (high dose); TCM-700C (low dose)
Drug: Placebo — Placebo, without acting ingredient.
  Other Names: Placebo, without acting ingredient.
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, multi-center, placebo controlled, three parallel arms, Phase IIb/III clinical study to evaluate the effects of adding a TCM-700C with a low or high dose onto the combination treatment (PegIFN plus RBV) for subjects with naive genotype 1 HCV infection.

This will be demonstrated by a higher sustained virologic response rate, defined as the absence of detectable HCV RNA 24 weeks after the termination of combination treatment, compared with the placebo add-on.

DETAILED DESCRIPTION:
Eligible subjects with written informed consent will be stratified according to their baseline HCV RNA (≤800,000 IU/mL versus>800,000 IU/mL), stage of liver fibrosis (METAVIR system fibrosis score of 0 1 versus 2 3).

During the 48 week Treatment Period and 24 week Follow up Period, subjects will be assessed at regular intervals for efficacy and safety at Weeks 2, 4, 8, 12, 16 and then every 8 weeks thereafter until study completion. If possible, subjects who prematurely discontinue the study during the Treatment Period will have samples taken for hematology, biochemistry and urinalysis in the same week of discontinuation as well as 24 weeks after discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects who are 20 to 65 years old (inclusive), of either gender and in any ethnical group in Asia.
* Chronic hepatitis C, positive with both antibody to hepatitis C virus (anti HCV) and HCV RNA assays.
* Confirmed HCV genotype 1.
* Subjects who are indicated to have combination treatment of PegIFNα 2a and RBV at the discretion of the investigator.
* All fertile males and females receiving RBV must be using two forms of effective contraception during treatment with study drugs and 6 months post treatment completion.
* Subjects must voluntarily give written informed consent indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Subjects must be able to comply with the assessments during the study.
* Subjects must be able to understand study QoL questionnaires.

Exclusion Criteria:

* Prior treatment with any IFN α or any medicines that contain Cordyceps.
* Prior treatment of hepatitis C with any other antiviral or immune modulators.
* Investigational therapy administered within 4 weeks, or within a time interval less than at least 5 half lives of the investigational agent, whichever is longer, prior to the first scheduled day of dosing in this study.
* Subjects diagnosed with hepatocellular carcinoma (HCC) by biopsy or α fetoprotein (AFP) serology and radiology (helical computed tomography [CT] and/or magnetic resonance imaging [MRI]) within 5 years of signing the informed consent form.
* Evidence of hepatic decompensation (history or current evidence of ascites, bleeding varices or hepatic encephalopathy).
* History or evidence of other liver diseases other than chronic HCV infection.
* Subjects with known allergy or hypersensitivity to any ingredient of the study drug or placebo.
* Pregnant, planning on becoming pregnant, or breastfeeding female subject or male subject whose partner is pregnant or planning on becoming pregnant.
* Subject with any of the following laboratory abnormalities:

  1. Platelet count <90,000/mm3;
  2. Absolute neutrophil count <1500 cells/mm3;
  3. Hemoglobin <12 g/dL for women and <13 g/dL for men;
  4. Creatinine >1.5 mg/dL;
  5. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >10 x upper limit of normal (ULN);
  6. Total serum bilirubin >1.5 x ULN;
  7. Subjects without cirrhosis and AFP >50 ng/mL must have an ultrasound between the screening and baseline visit with no findings suspicious for HCC.
* Medical conditions which are contraindications for PegIFNα 2a or RBV therapy:

  1. Psychiatric disorders;
  2. Organ transplant (other than cornea or hair transplant or skin graft);
  3. Severe concurrent medical disease such as severe hypertension, significant coronary heart disease, poorly controlled diabetes mellitus (glycated hemoglobin A1c [HbA1c] >8.5%), not adequately controlled thyroid dysfunction, chronic obstructive pulmonary disease, severe infections (bacterial, viral, fungal, including acute tuberculosis), or hemoglobinopathies (thalassemia major or sickle cell anemia);
  4. Autoimmune hepatitis or other autoimmune conditions known to be exacerbated by PegIFNα 2a and RBV.
* History of a severe seizure disorder or current anticonvulsant use.
* Evidence of severe retinopathy (e.g., cytomegalovirus retinitis, macular degeneration) or clinically relevant ophthalmological disorder (e.g., due to diabetes mellitus or hypertension).
* Other cases judged by the investigator to be ineligible for participation in the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2018-03 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
sustained virologic response (SVR) rate | 24 weeks after the end of treatment (EOT, 48 weeks)
  undetectable HCV RNA 24 weeks after the EOT.

SECONDARY OUTCOMES:
Virologic response (VR) | at the EOT (48 weeks)
  undetectable HCV RNA at the EOT.
relapse rate | 24 weeks after the EOT
  undetectable HCV RNA at the EOT followed by a positive HCV RNA level within 24 weeks after the EOT

CONTACTS AND LOCATIONS:
Overall Officials: I-Shyan Sheen, MD, Principal Investigator — Chang Gung Memorial Hospital; Lai Wei, MD, Principal Investigator — Peking University People's Hospital
Locations (2):
- Peking University People's Hospit, Beijing, Beijing Municipality, China
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No